CLINICAL TRIAL: NCT00199160
Title: Efficacy and Activity of BAY 43-9006 in Patients With Recurrent and/or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAY 43-9006 Head and Neck
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2005-09

CONDITIONS: Head and Neck Neoplasms
Keywords: local recurrence and or metastatic disease; Previously treated with platinum; carcinoma of the head and neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Sorafenib

INTERVENTIONS:
Drug: BAY 43-9006

SUMMARY:
This is a Phase II trial evaluating the efficacy and the biological activity of BAY 43-9006 in patients with recurrent and/or metastatic head and neck cancer.

DETAILED DESCRIPTION:
This is a Phase II trial evaluating the efficacy and the biological activity of BAY 43-9006 in patients with recurrent and/or metastatic head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients (18 years old and above), with a histologically proven, measurable, locally recurrent, and/or metastatic head and neck tumor.
* > 4 weeks since major surgery
* > 4 weeks since prior chemotherapy
* > 3 weeks since prior therapy with biological agents (Interleukin-2 [IL-2], interferon, other molecular-targeted therapies [except Ras/Raf inhibitors]).
* Performance status < 2
* Life expectancy > 3 months.
* At least one uni-dimensional measurable lesion by computed tomography (CT)-scan or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Adequate liver, pancreatic, renal, and coagulation function
* A slide or paraffin-block from a tumor biopsy MUST be available at the time of screening. If the original diagnostic biopsy is not available at the time of screening, an additional biopsy is required.

Exclusion Criteria:

* Severe preexisting conditions
* Evidence of bone marrow suppression
* Frequent vomiting or medical condition, which could interfere with oral medication intake
* Lack of resolution of all toxic manifestations of prior chemotherapy, biologic, or radiation therapy (alopecia excluded).
* Known HIV positivity or AIDS-related illness.
* Previous exposure to a Ras/Raf inhibitor
* Previous malignancy (except for cervical carcinoma in situ, adequately treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis and T1] or other malignancies curatively treated > 2 years prior to entry)
* Congestive heart failure
* Cardiac arrhythmias requiring anti-arrhythmics
* Active coronary artery disease or ischaemia
* Active clinically serious bacterial or fungal infections
* Known brain or meningeal metastases
* Patients with seizure disorder requiring medication (such as anti-epileptics)
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test.
* Concurrent anti-cancer chemotherapy or immunotherapy is excluded
* Significant surgery within four weeks prior to start of study drug
* Investigational drug therapy outside of this trial, or any chemotherapy during or within 4 weeks prior to start of study drug
* Myelosuppressive radiotherapy within four weeks prior to start of study drug (short-course non-myelosuppressive radiotherapy may be allowed based on approval of principal investigators)
* Concomitant treatment with ketoconazole, itraconazole, ritonavir, or use of grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
PFS

CONTACTS AND LOCATIONS:
Overall Officials: AHMAD AWADA, Principal Investigator — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium